CLINICAL TRIAL: NCT05989984
Title: Monocentric, Prospective, Randomized Study to Evaluate the Efficacy of a New Iron Supplement with Orodispersible Formulation Vs an Iron Supplement in Capsules in Subjects with Mild Anemia
Brief Title: Efficacy Evaluation of an ODF Iron Supplement Vs an Iron Supplement in Capsules in Subjects with Mild Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IBSA Farmaceutici Italia Srl (Industry)
Collaborators: Informapro Srl (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IBSAFE_CLI22
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Iron Deficiencies
MeSH Terms: conditions — Iron Deficiencies | interventions — Iron-Dextran Complex; Capsules; sucrosomial iron

STUDY DESIGN:
Intervention Model Description: Monocentric, prospective, randomized study
Masking Description: No masking procedure will be applied
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ODF Iron Supplement (Experimental): ODF iron supplement contains 30 mg of elemental iron (corresponding to 120 mg of ferric pyrophosphate) and 400 μg of folic acid.
  Interventions: Dietary Supplement: ODF Iron Supplement
- Iron Supplement in Capsule (Active Comparator): Iron supplement in capsule contains 30 mg of elemental iron (corresponding to 120 mg of ferric pyrophosphate) and 70 mg of vitamin C.
  Interventions: Dietary Supplement: Iron Supplement in Capsules

INTERVENTIONS:
Dietary Supplement: ODF Iron Supplement — ODF iron supplement will be admistered daily for 8 weeks.
  Arms: ODF Iron Supplement
Dietary Supplement: Iron Supplement in Capsules — Iron supplement in capsule will be admistered daily for 8 weeks.
  Other Names: Sucrosomial iron
  Arms: Iron Supplement in Capsule

SUMMARY:
The aim of the study is to evaluate the efficacy of a new iron supplement with orodispersible formulation vs an iron supplement in capsules in subjects with mild anemia.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the efficacy of a new iron supplement with orodispersible formulation in modulating peripheral blood biomarkers of iron levels in subjects with mild anemia after 8 weeks of supplementation, compared to baseline values and also aims to evaluate its acceptability. For the evaluation, an iron supplement in capsules will be used as a comparison supplement.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent signed prior to inclusion in the study
* 18-55 years
* Ability to understand the nature and the purpose of the study, including possible risks and side effects
* Capability to collaborate with the investigator and meet the requirements of the entire study
* Subjects with mild anemia (with WHO hemoglobin values between 11-11.9 g/dl for women and between 11-12.9 g/dl for men)

Exclusion Criteria:

* Clinically significant abnormalities in the ECG evaluation
* Clinically significant abnormal laboratory values indicative of disease
* Known allergy or presumed hypersensitivity to the food supplement investigated (iron) and / or to the excipients of the two formulations
* History of anaphylaxis from drugs, dietary supplements or allergic reactions in general, which the investigator believed could influence the outcome of the study
* Significant history of kidney, liver, gastrointestinal, cardiovascular, respiratory, skin, haematological, endocrine or neurological diseases that may interfere with the purpose of the study
* Taking herbal remedies and dietary supplements (including iron supplements, supplements with vitamin C, supplements with folic acid, supplements with vitamin B12, multivitamins) in the 2 weeks prior to the start of the study
* Taking corticosteroids, thyroid hormones, antibiotics, antiepileptics
* Alcohol abuse
* Any clinical condition that in the investigator's judgment is deemed incompatible with study participation
* Women who are pregnant or breastfeeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2023-07-29 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in blood concentration of hemoglobin with ODF iron supplement (test product) | Day 0, Week 8
  Change from baseline in blood concentration of hemoglobin after 8 weeks of supplementation with ODF iron supplement

SECONDARY OUTCOMES:
Change from baseline in blood concentration of hemoglobin with test product | Day 0, Week 4
  Change from baseline in blood concentration of hemoglobin after 4 weeks of supplementation with test product
Change from baseline in blood concentration of hemoglobin with Iron supplement in capsule (reference product) | Day 0, Week4, Week 8
  Change from baseline in blood concentration of hemoglobin after 8 weeks of supplementation with Iron supplement in capsule
Change from baseline in blood concentration of hematocrit | Day 0, Week4, Week 8
  Evalution of the change from baseline of hematocrit after administration of test versus reference product
Change from baseline in blood concentration of ferritin | Day 0, Week4, Week 8
  Evalution of the change from baseline of ferritin after administration of test versus reference product
Change from baseline in blood concentration of transferrin | Day 0, Week4, Week 8
  Evalution of the change from baseline of transferrin after administration of test versus reference product
Change from baseline in blood concentration of transferrin receptor | Day 0, Week4, Week 8
  Evalution of the change from baseline of transferrin receptor after administration of test versus reference product
Change from baseline in blood concentration of folic acid | Day 0, Week4, Week 8
  Evalution of the change from baseline of folic acid after administration of test versus reference product
Change from baseline in blood concentration of serum iron | Day 0, Week4, Week 8
  Evalution of the change from baseline of serum iron after administration of test versus reference product
Change from baseline in mean corpuscolar volume (MCV) | Day 0, Week4, Week 8
  Evalution of the change from baseline of MCV after administration of test versus reference product

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Angeletti, Principal Investigator — Operative Research Unit of Clinical Laboratory
Locations (1):
- Fondazione Policlinico Universitario Campus Bio-Medico di Roma, Roma, Italy, Italy